CLINICAL TRIAL: NCT06879756
Title: Relationship Between Flexible Flat Foot and Lumbar Proprioception
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Anwar Mohamed Elmeligy, principal investigator, Cairo University
Other Study IDs: Hoda-005289
Record Dates: First submitted 2025-03-10; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Flexible Flatfoot; Lumbar Spine Injury; Proprioceptive Disorders
MeSH Terms: conditions — Flatfoot; Spinal Injuries; Somatosensory Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- flexible flat feet: 28 patients suffering from flexible flatfoot were included in this group
- normal subjects: 27 normal subjects were included in this group

SUMMARY:
The purpose of this study was to determine the relationship between flexible flatfoot and lumbar proprioception.

DETAILED DESCRIPTION:
The human foot plays a crucial role in maintaining balance during various activities, and poor foot alignment, such as excessive subtalar joint pronation, can lead to leg, knee, and back pain. Proprioception is essential for active joint stability, as it indirectly modulates and provides motor response, helping the neuromuscular system maintain balance. Lumbar proprioception deficits can decrease the ability to assume a neutral spinal posture and coordinate muscle contraction, affecting spinal segmental function, dynamic joint stability, and good motor control. This study investigates the association between flatfoot and lumbar proprioception.

ELIGIBILITY:
Inclusion Criteria:

* 60 subjects of both sexes (females and males) were selected and assigned into two groups
* Patient's age range was between 17 to 30 years old.
* Subjects with flexible flat foot posture according to the Navicular Drop Test by Brody method: a normal foot (between five and nine mm of navicular drop), pronated foot (more than 10 mm of navicular drop).
* Patients will be willing and able to participate in assessment without cognitive impairments that would limit their participation

Exclusion Criteria:

The potential participation was excluded when they had one of the following criteria:

* Repeated lower extremity injuries, such as fractures or deformities.
* History of surgery to the lower extremity.
* history of back surgery
* rheumatologic disorders
* spine infections
* ankle fracture
* lumbar fracture
* spondylosis
* lumbar disc bulge
* spondylolisthesis

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: • Subjects with flexible flat foot posture according to the Navicular Drop Test by Brody method: a normal foot (between five and nine mm of navicular drop), apronated foot (more than 10 mm of navicular drop).
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
assessment of the foot posture using navicular drop test | at baseline
  The study evaluates foot posture in a weight-bearing position by placing the thumb and index fingers on the medial and lateral aspects of the talar dome. The subject is then asked to invert and evert the hind-foot and ankle until equal depressions are felt. The distance between the navicular tubercle and the floor is measured. The navicular-drop score is recorded, and the subject is classified into a pronated foot (more than 10 mm of navicular drop) and a normal foot (between five and nine mm of navicular drop).

SECONDARY OUTCOMES:
assessment of change of lumbar proprioception using Biodex system isokinetic dynamometer | at baseline
  The Biodex System 3 Pro isokinetic device is used to measure lumbar proprioception. The device offers isokinetic, eccentric, isometric, and passive modes for all body joints and is equipped with various attachments and isolation straps. The system is equipped with a computer unit and a special testing unit for lumbar area testing. Subjects are instructed to sit on the lumbar attachment unit with their hips and knees flexed at 90 degrees, strapped around their thigh, pelvis, and trunk, and fold their arms above their chest. The selected test is active repositioning error/speed 30o/S, with a target position of 30° lumbar flexion. The device is locked in 0° position during trials, and the isokinetic device software calculates the mean of the three real testing results. The isokinetic machine prints the results, providing each trial's error value and the average error of the three trials.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No